CLINICAL TRIAL: NCT02458001
Title: Developing a Stepped Approach to Improving Sexual Function After Gynaecological Cancer- a Feasibility Study and Randomized Controlled Trial
Brief Title: Developing a Stepped Approach to Improving Sexual Function aFteR Treatment fOr gyNaecological Cancer
Acronym: SAFFRON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA 11/111/02
Record Dates: First submitted 2015-03-20; First posted 2015-05-29 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Cervical Cancer; Ovarian Cancer; Uterine Cancer; Vaginal Cancer; Vulval Cancer; Psychosexual Dysfunctions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAFFRON stepped care (Experimental): 3 level intervention: level 1:Self help booklet level 2: CNS delivered intervention level 3: psychologist delivered intervention
  Interventions: Behavioral: SAFFRON stepped care
- enhanced treatment as usual (ETU) (No Intervention): level 1 intervention: self help booklet Non study trained CNS will offer assessment, advice, vaginal dilator training where appropriate, arrange topical oestrogens or other creams

INTERVENTIONS:
Behavioral: SAFFRON stepped care — Behavioral: SAFFRON stepped care Stepped care (Improving Access to Psychological Therapies, 2012; Richards et al., 2012) adapted for the gynaecological cancer setting to produce a 3-step model including a clinical assessment and treatment algorithm.
  Assessment Algorithm FSFI Interventions
  Level 1:
  Best available self-help literature on psychosexual difficulties after cancer as judged by the project team and two patient advocates.
  Level 2:
  A 3-5 session manualised psycho-educational intervention delivered fortnightly by study trained CNSs with taping and supervision for adherence to protocol and manual.
  Level 3:
  16 weekly session manualised brief psychotherapy adaptation of InterPersonal Therapy, IPT (Interpersonal Psychotherapy for Sexual Adjustment post Gynaecological Cancer, IPT-APGyC)
  Arms: SAFFRON stepped care

SUMMARY:
Women affected by gynaecologic cancers are often not aware of sexual consequences of cancer and its treatment. Most do not receive appropriate advice or help to recover sexual function, and the impact on their sexuality may be profound. Despite this several potential therapies can be effective in helping recovery. A major challenge is informing and involving the patients in an appropriate and sensitive manner, and a further issue is the delivery of such therapies in busy and medically driven gynaecologic oncology clinics. It will use and adapt existing evidence based therapies for improving sexual function after cancer treatment and develop a model for delivering these in the NHS (United Kingdom National Health Service) setting. The model of 'stepped care' is adapted from that used nationally and successfully in the Increasing Access to Psychological Therapies (IAPT) programme. Assessment allows for 'stepping up and down', i.e. calibrating the type of help a woman receives according to need and her response to treatment already given.This study will develop and evaluate a 'stepped' system of interventions using elements of best available evidence, adapting existing interventions to help women recover their sexual feelings and activity, starting with simple methods, moving on to new talking treatments for more complex cases. The investigators address all gynaecologic cancers on the principle that sexual difficulty is the problem the investigators are treating, not the cancer of origin. Ongoing clinical assessment will be vital for the success of the stepped care model. The investigators will deliver training and supervision to enhance the skills needed by the Clinical Nursing Specialist (CNS). An important part of this study will be characterising the range of women and their willingness to participate in psychosexual help. One-to-one follow up interviews will inform the level of input required for any subsequent Randomised Control Trial (RCT). The investigators will use internationally recognised rating scales for rating sexual function, assess how illness and treatment affect mood and self esteem. The investigators will also measure the overall cost-effectiveness to the public sector of providing this treatment, compared to costs of subsequent use of health and social services. This pilot study will assess the feasibility of conducting a full scale investigation of a stepped therapy and indicate the potential benefits to the patients, their partners, and to the NHS generally.

DETAILED DESCRIPTION:
Many cancer patients have sexual difficulties , gynaecologic cancer (Gyn-Onc) patients are particularly vulnerable to changes in sexual activity and lack of sexual desire with sexual difficulty rates estimated between 40 and 100% . Women undergo a range of treatments for ovarian, cervix, womb and vulval cancer with different combinations of surgery, chemotherapy, and radiation. Some treatments have a deleterious effect on women's internal and external sex organs, surrounding tissues and nerves, and render some menopausal. Following such treatments women report a wide range of difficulties including loss of libido, dyspareunia, vaginal dryness, and orgasmic difficulty. In addition, the symptom burden of gynaecologic cancers is heavy with many women reporting pain, fatigue, changes in bowel function, urinary symptoms including leakage, and depression and anxiety which interact with menopausal and sexual difficulties. The major impact of physical well-being on sexual function has been noted, as well as the lack of relationship between extent of treatment and formal scores of sexual function. Unsurprisingly, women treated for gynaecologic cancer are at high risk of emotional distress. One prevalence study found 23% satisfying criteria for major depressive disorder and another found greater depressive symptoms in gyn-onc patients than in breast, urology or gastro intestinal cancers. It is suggested that some of the depressive symptoms are related to the very high levels of sexual difficulty experienced after treatment. Some suggest that sexual self schema is an important moderator of response, finding positive sexual self schema associated with more frequent sexual activity, better sexual responsiveness, and higher global sexual satisfaction across all disease sites and confounders, suggesting it makes women more resilient to the adverse sexual impacts of gynaecologic cancer. Despite their sexual difficulties, many gynaecologic cancer survivors resume intercourse. Frequency of intercourse in one sample was comparable to available norms for similarly aged women, but these and other longitudinal data have shown sexual satisfaction and responsiveness significantly impaired following treatment. Patients report sexuality rarely addressed by physicians. It has been found that conversation with physicians about sexual effects of cancer is associated with significantly lower likelihood of complex sexual morbidity among very long-term survivors; but 62% of 221 participants reported their physician had never initiated a discussion about sexuality after cancer. Examining sexuality in palliative care, it has been found that patients consider it important to talk about sexuality and to face it with an experienced professional even though life expectancy is short. Patients in that study had not had this opportunity. Moreover, some patients were still able to maintain a sufficient sexual activity, in terms of quality and quantity.Nursing researchers found that cancer nurses were more likely to focus on the technical aspects of sexual recovery post treatment, for example vaginal dilation, and offered minimal advice or opportunities for disclosure for sexual dysfunctions, dissatisfaction with partner relationships or mood and other psychological difficulties. Clinical Nurse Specialists (CNSs) in gynaecologic cancer acknowledge that they have an important role in this aspect of care but do not always feel confident or competent to assess or manage patients psycho-sexual needs, and appropriate referral is then problematic . A recent review of specific complaints of all cancer patient referrals to the Sexual Health Program of the Memorial Sloan Kettering Cancer Center found that most sought help for painful intercourse (65%), vaginal dryness (63%), low sexual desire (46%), and orgasmic disorder (7%). The first two of these are partially managed through current best treatment, i.e. topical estrogen, vaginal dilators and lubricants. Prevalence reports by cancer site include a comparison of crude prevalence (66.67%) with age-standardized prevalence (55%) in cervical cancer. Many other studies report ranges from 83% sexual difficulties, to 66% significant and 46% moderate difficulties. In early stage cervix cancer treated with radical hysterectomy, 65.8% were reported to have sexual difficulties. In contrast with most sexual therapy interventions where anxiety reduction is often key, management of low sexual desire in the context of gynaecologic cancer requires an intervention which additionally addresses the wider range of mediating factors, including loss, life-threat, trauma, change of body image, pre-existing psychological outlook, mood, depression and anxiety symptoms as well as the relationship within which the woman finds herself. A wide range of non-controlled trials of sexual therapy interventions are reported in reviews across a range of interventions. All show small effect sizes, but are accompanied by patient satisfaction. A Cochrane Review of RCTs for psycho-sexual dysfunction in women treated for gynaecologic cancer concluded, 'there is insufficient evidence to support or refute the use of any interventions for psychosexual dysfunction after gynaecologic cancer.' Further, they suggested that future trials required multi-center RCTs with outcome measures validated in gynaecologic cancer patients. 'When considering interventions to trial, the investigators would suggest that investigators should focus on interventions that can be delivered by existing members of the multidisciplinary team treating women with gynaecologic cancers. It is more likely that such measures, if found effective, will be affordable and capable of being integrated into standard care. An international consensus on outcome measures would greatly facilitate the comparison of interventions in the future.' This study attempts to address this for the NHS by using the existing multi-disciplinary team to deliver a stepped care approach. This involves CNS delivered interventions at step 1 and step 2 as the major treatment delivery, and only a small minority of more complex psychological issues being treated at step 3 by a level 4 practitioner to whom patients should have access according to peer review.From the evidence above, it is often the case that women affected by gynaecologic cancer are not aware of basic information about the sexual consequences of their gynaecologic cancer and its treatment, and do not receive appropriate advice or help to recover sexual function, and adapt to their changed body and relationships. It is generally recognized by two Cochrane reviews that new interventions are needed for sexual dysfunction in gynaecological cancer and these need to be examined in multi-center RCTs with agreed outcome measures. There is a sizable population with these problems to be addressed as there are currently 1.8 million people in England living with and beyond cancer, and 2 million across the UK as a whole. This number is likely to grow by over 3% per year, reflecting the increasing incidence of cancer and better survival rates. By 2030 there are likely to be around 3 million cancer survivors in England. Since the investigators have the ability to develop suitable treatments, the investigators have a duty to explore them. The current acceptance of the worth of well-being, and conversely the cost of depression, anxiety or unwillingness to engage with the healthcare system - all potential long term effects for the patient group concerned - are drivers for this research. Better awareness of mental health issues and depression in general and in cancer patients plus greater acceptance that these symptoms have causes which can be treated or addressed is relevant too. In addition the work is planned at a time when there is more awareness of sexual health, and evidence from cancer user groups, policy makers) and research of more openness to discuss these matters as a medical need. The potential of CNSs to deliver interventions to help with the consequences of cancer treatment has been recognized by the UK Department of Health yet little is known about CNS's training or supervisory needs to provide interventions for psycho-sexual dysfunction to work alongside psychologists. If care pathways exist for addressing sexual dysfunction in cancer they are currently unique to individual units; providing the evidence for pathways which better meet the requirements of the population will facilitate clinical application of more appropriate and consistent practice. What is needed is a study to develop interventions and test them to facilitate best practice in treatment of sexual dysfunction for all relevant women in gynaecologic cancer centres.

Trial objectives:Aims: To establish whether women treated for gynaecologic cancer with moderate to severe sexual dysfunction are willing to participate in a randomized trial model and adhere to treatment 1)To indicate likely rates of recruitment to a future evaluation of the SAFFRON intervention2)To pilot a stepped care psycho-sexual intervention (SAFFRON) on the IAPT model3)To establish whether the SAFFRON intervention is acceptable to patients4)To establish whether SAFFRON is deliverable by a Gyn-Onc cancer center multidisciplinary team;5)To indicate the most appropriate outcome measures for use in a larger trial6)To inform estimates of the likely effect size, which will assist sample size calculations for a larger trial Research questions:To establish whether women treated for gynaecological cancer with moderate to severe sexual dysfunction are willing to participate in a randomized trial model and adhere to treatment

1. Will women agree to be randomized to a sexuality intervention?
2. Are different tumor sites, treatments, cancer stages at approach associated with different rates of uptake of therapy/intervention of recruitment to trial?
3. Is stepped care operable within the NHS system as it stands?
4. What is the likely effect of three levels of intervention on sexual function, mood and self-esteem as measured by standard measures?
5. What is the rate of attrition from each treatment modality? Purpose of Research a)Is it possible to improve sexual functioning for women treated for gynaecological cancer within the current clinical setting of NHS gynaecological cancer treatment?b)Can a suitable intervention be developed and evaluated in a feasibility trial?c)Can a suitable intervention be developed and evaluated in a feasibility trial?d)Is a stepped approach acceptable and practical?e)Can it be done within NHS settings?

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 (with partners at their choice) treated for any gynaecological malignancy with surgery and/or chemotherapy and/or radiation at UCLH (University College London Hospitals) Gynaecological Cancer Centre or University Hospitals Bristol Gynaecological Cancer Centre
* 3 months minimum post end of treatment
* any sexual orientation
* with sexual function difficulties identified by initial screen (3 clinical questions within clinical interview posed by doctor or nurse)

Exclusion Criteria:

* Poor English
* Current drug or alcohol abuse
* Current sexual therapy or psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 24 months
  measure of feasibility
Consent rate to randomization and treatment | 24 months
  measure of feasibility
Proportion of women stepping up from level 1 to 2, and level 2 to 3 | 24 months
  measure of feasibility
Proportion of women dropping out of therapy | 24 months
  measure of feasibility
Number of usable data points from all measures at all time points | 24 months
  measure of feasibility
Proportion of women lost to follow-up on trial measures | 24 months
  measure of feasibility

SECONDARY OUTCOMES:
Change in Female Sexual Function Index (FSFI) | 24 months
  shows whether interventions have changed sexual functioning

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Gessler, PhD, Principal Investigator — University College, London

REFERENCES:
- [Derived] Gessler S, King M, Lemma A, Barber J, Jones L, Dunning S, Madden V, Pilling S, Hunter R, Fonagy P, Summerville K, MacDonald N, Olaitan A, Lanceley A. Stepped approach to improving sexual function after gynaecological cancer: the SAFFRON feasibility RCT. Health Technol Assess. 2019 Feb;23(6):1-92. doi: 10.3310/hta23060. PMID 30798790